CLINICAL TRIAL: NCT05008978
Title: The Effects on Glycemic and Insulinemic Responses by Fruit Consumption (TGIF Study)
Brief Title: The Effects on Glycemic and Insulinemic Responses by Fruit Consumption
Acronym: TGIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019/00691
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: time effects on fruit consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test 1 (Experimental)
  Interventions: Other: Test 1
- Test 2 (Experimental)
  Interventions: Other: Test 2
- Test 3 (Experimental)
  Interventions: Other: Test 3
- Test 4 (Experimental)
  Interventions: Other: Test 4
- Test 5 (Experimental)
  Interventions: Other: Test 5

INTERVENTIONS:
Other: Test 1 — 25g of available carbohydrates from White bread with 25g of available carbohydrates from Banana consumed simultaneously at time 0 min
  Arms: Test 1
Other: Test 2 — 25g of available carbohydrates from Banana consumed at time -15 min and 25g of available carbohydrates from white bread consumed at time 0 min
  Arms: Test 2
Other: Test 3 — 25g of available carbohydrates from White bread consumed at time 0 min and 25g of available carbohydrates from Banana consumed at time 15 min
  Arms: Test 3
Other: Test 4 — 25g of available carbohydrates from White bread with 25g of available carbohydrates from Papaya consumed simultaneously at time 0 min
  Arms: Test 4
Other: Test 5 — 25g of available carbohydrates from White bread with 25g of available carbohydrates from Apple consumed simultaneously at time 0 min
  Arms: Test 5

SUMMARY:
The health benefits of fruits and their importance in a healthy diet have long been known. Several intervention studies have included the promotion of fruit as part of the healthy diet and epidemiologic evidences have demonstrated that a diet rich in fruits is associated with the reduction in the risk of many chronic diseases, including type 2 diabetes. Such beneficial health effects of fruits could be attributed to the presence of dietary fiber, micronutrients (vitamins and minerals), antioxidants and phytochemicals found in them. However, up to our knowledge, no study has investigate the time-course effects on the co-ingestion of fruits with other food product on postprandial glycaemic response (GR) and insulinaemic response (IR). The time-course effect will be examined in this study in order to determine its optimal effect on GR and IR. The investigators also aimed to compare the effects of varying micronutrients content in fruits on GR and IR.

DETAILED DESCRIPTION:
Type 2 diabetes is one of the most common non-communicable diseases found in 415 million adults worldwide in 2015 and the number is expected to increase to 642 million in 2040. This has serious consequences for healthcare expenditure as it has been estimated that the global health expenditure on diabetes is at least USD$673 billion in 2015 and is forecasted to increase to USD$802 billion in 2040. This creates a major public health burden and effective treatments and prevention strategies are necessary. The Asian phenotype has been shown to be more susceptible to diabetes compared to the Western phenotype where more than half (56%) of the population with type 2 diabetes lived in the South-East Asia Region or the Western Pacific Region in 2015.Pharmacological methods through the use of drugs and insulin remains as the conventional strategy in the management of type 2 diabetes. However, in recent years, dietary interventions have been used as a mean to prevent or delay the onset of type 2 diabetes. Food has now become the new medicine and a healthy diet is widely believed to play an important role in the prevention of the development of type 2 diabetes.The health benefits of fruits and their importance in a healthy diet have long been established. Several intervention studies have included the promotion of fruit as part of the healthy diet with epidemiological evidences demonstrating that a diet rich in fruits is associated with a reduction in the risk of many chronic diseases, including type 2 diabetes. Such beneficial health effects of fruits may be attributed to the presence of dietary fibre, micronutrients (vitamins and minerals), antioxidants and phytochemicals found in them. However, to our knowledge, no study has investigated the time-course effects of co-ingesting fruits with a carbohydrate-based food product on postprandial glycaemic response (GR) and insulinaemic response (IR). GR and IR is the effect a food product has on blood glucose and insulin levels respectively, after consumption. Better control of GR and IR were found to be associated with a lower risk of development of type 2 diabetes and other cardiovascular diseases. Studies have shown that soluble dietary fibre, which are found in fruits, decrease the rise in blood glucose and insulin level. Addition of fibre as a food ingredient was also found to modulate glucose response by improving insulin sensitivity. Antioxidants and phytochemicals in fruits have also been hypothesized to improve insulin sensitivity and hence protect against diabetes. In the second part of the study, the investigators aim to compare the effects of varying micronutrients content in fruits on GR and IR. Fruits have highly variable contents of fibre, antioxidants, other nutrients, and phytochemicals that may jointly influence the risk of metabolic diseases. It has been reported that the consumption of higher anthocyanins content had an inverse relationship with the risk of developing type 2 diabetes. Varying content of resveratrol, chlorogenic acid and naringin have also been reported to have an association with the risk of type 2 diabetes in animal studies. Due to the heterogeneous composition found in fruits, it may be plausible that different fruits have varying effects on GR and IR. Therefore, the investigators hypothesized that varying micronutrients content in fruit plays an essential role in the association with diabetes risk due to a difference in GR and IR. In this proposed study, the investigators will thus determine whether different micronutrients content present in different fruits have an effect on postprandial on GR and IR.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese Ethnicity
* Age between 21-50 years
* Weight of at least 45 kg
* Body mass index between 18.5 - 25 kg/m2 (inclusive)
* Fasting blood glucose < 5.6 mmol/L
* Normal blood pressure ≤140/90 mmHg

Exclusion Criteria:

* People who smoke
* People with any metabolic diseases or cardiovascular diseases (such as heart disease, hypertension, diabetes mellitus, etc.)
* Having any other diseases involving the small intestine or the colon (e.g., irritable bowel syndrome, inflammatory bowel disease, gastric reflux) or having any liver or kidney disorders or any family history of kidney stones
* People with known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
* People taking any prescribed medication or dietary supplements which may interfere with the study measurements
* People with medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Individuals who have any major organ dysfunction (e.g. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* Individuals who have any known food allergies to the food components of the study protocol
* People who intentionally restrict food intake
* Individuals who partake in sports at the competitive and/or endurance levels
* People having active Tuberculosis (TB) or currently receiving treatment for TB
* People who have any known chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* People who are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Have known history of anaemia or thalassemia minor
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC
* Participants who are found to be repeatedly difficult to cannulate

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All healthy male subjects
Enrollment: 15 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose | 180min
  Baseline venous blood was collected by cannulation into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA. Analyse using Beckman Coulter analyser. (time frame 180min)

SECONDARY OUTCOMES:
Differences in postprandial glycaemic response among banana, papaya and apple | 180min
  Baseline venous blood was collected by cannulation into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA. Analyse using Beckman Coulter analyser. (time frame 180min)
Differences in insulinaemic response among banana, papaya and apple | 180min
  Baseline venous blood was collected by cannulation into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA. Analyse using Beckman Coulter analyser. (time frame 180min)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No